CLINICAL TRIAL: NCT04586231
Title: An Open-label, Randomized, Phase 3 Study of MK-6482 in Combination With Lenvatinib (MK-7902) vs Cabozantinib in Participants With Advanced Renal Cell Carcinoma Who Have Progressed After Prior Anti-PD-1/L1 Therapy
Brief Title: A Study of Belzutifan (MK-6482) in Combination With Lenvatinib Versus Cabozantinib for Treatment of Renal Cell Carcinoma (MK-6482-011)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-011; MK-6482-011 (Other: MSD); jRCT2031210311 (Other: jRCT(Japan Registry of Clinical Trials)); 2024-510620-39 (Registry Identifier: EU CT); U1111-1302-2815 (Registry Identifier: UTN); 2020-002075-35 (EudraCT Number)
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — belzutifan; lenvatinib; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belzutifan + Lenvatinib (Experimental): Belzutifan 120 mg and lenvatinib 20 mg orally once a day
  Interventions: Drug: Belzutifan; Drug: Lenvatinib
- Cabozantinib (Active Comparator): Cabozantinib 60 mg orally once a day
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Belzutifan — Immediate-release 40 mg tablet
  Other Names: PT2977; MK-6482; WELIREG™
  Arms: Belzutifan + Lenvatinib
Drug: Lenvatinib — Capsule available in 4 mg and 10 mg dosages
  Other Names: Lenvima; E7080; MK-7902
  Arms: Belzutifan + Lenvatinib
Drug: Cabozantinib — Tablet available in 20 mg, 40 mg and 60 mg dosages
  Other Names: Cabometyx; Cometriq; XL184; BMS-907351
  Arms: Cabozantinib

SUMMARY:
This study will compare the efficacy and safety of belzutifan + lenvatinib versus cabozantinib in participants with advanced renal cell carcinoma (RCC) with clear cell component after prior therapy.

The primary hypothesis is that belzutifan + lenvatinib is superior to cabozantinib in terms of progression-free survival or overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, locally advanced or metastatic clear cell renal cell carcinoma (RCC).
* Disease progression on or after an anti-programmed cell death-1/ligand 1 (PD-1/L1) therapy as either first or second-line treatment for locally advanced/metastatic RCC or as adjuvant treatment or neoadjuvant/adjuvant with progression on or within 6 months of last dose.
* Measurable disease per RECIST 1.1 criteria as assessed by local study investigator.
* Karnofsky performance status (KPS) score of at least 70% assessed within 10 days before randomization.
* Received no more than 2 prior systemic regimens including: one anti-PD-1/L1 containing adjuvant or neoadjuvant/adjuvant regimens with progression on or within 6 months from the last dose of that regimen OR one or 2 regimens for locoregional/advanced disease
* Received only 1 prior antiPD-1/L1 therapy for adjuvant, neoadjuvant/adjuvant or locally advanced/metastatic RCC.
* A male participant is eligible to participate if he is abstinent from heterosexual intercourse or agrees to use contraception during the intervention period and for at least 7 days after the last dose of belzutifan or lenvatinib in the belzutifan+lenvatinib arm, whichever occurs last, and 23 days after the last dose of cabozantinib.
* A female participant is eligible to participate if they are not pregnant, not breastfeeding, and at least 1 of the following conditions applies: Not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the intervention period and for at least 30 days after the last dose of study intervention in the belzutifan+ lenvatinib arm, or 120 days after the last dose of study intervention in the cabozantinib arm.
* Adequately controlled blood pressure.
* Adequate organ function.

Exclusion Criteria:

* A pulse oximeter reading <92% at rest, requires intermittent supplemental oxygen, or requires chronic supplemental oxygen.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy.
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Clinically significant cardiac disease within 6 months of first dose of study intervention.
* Prolongation of QTc interval to >480 ms.
* Symptomatic pleural effusion (e.g.,cough, dyspnea, pleuritic chest pain) that is not clinically stable.
* Pre-existing ≥Grade 3 gastrointestinal or nongastrointestinal fistula.
* Moderate to severe hepatic impairment.
* History of significant bleeding within 3 months before randomization.
* History of solid organ transplantation.
* Known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.
* Unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (e.g., gastrectomy, partial bowel obstruction, malabsorption).
* Known hypersensitivity or allergy to the active pharmaceutical ingredients or any component of the study intervention formulations.
* Received colony-stimulating factors [eg, granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GMCSF) or recombinant erythropoietin (EPO)] within 28 days before randomization.
* Prior treatment with belzutifan or another hypoxia-inducible factor (HIF)-2α inhibitor.
* Prior treatment with lenvatinib.
* Prior treatment with cabozantinib.
* Currently participating in a study of an investigational agent or using an investigational device.
* Active infection requiring systemic therapy.
* History of human immunodeficiency virus (HIV) infection.
* History of hepatitis B or known active hepatitis C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2027-02-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 34 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review will be presented.
Overall Survival (OS) | Up to approximately 44 months
  OS is defined as time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 24 months
  ORR is defined as the percentage of participants who have a complete response (CR: Disappearance of all target lesions) or a partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR as assessed by blinded independent central review based on RECIST 1.1 will be presented.
Duration of Response (DOR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 44 months
  For participants who demonstrate a confirmed complete response (CR: Disappearance of all target lesions) or confirmed partial response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death. The DOR as assessed by blinded independent central review will be presented.
Number of Participants Who Experienced One or More Adverse Events (AEs) | Up to approximately 44 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE) | Up to approximately 44 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (184):
- United States (33):
  - Ironwood Cancer & Research Centers ( Site 0077), Chandler, Arizona
  - Cedars Sinai Medical Center ( Site 0027), Los Angeles, California
  - UCLA Hematology/Oncology - Santa Monica ( Site 0048), Los Angeles, California
  - St. Joseph Hospital-The Center for Cancer Prevention and Treatment ( Site 0095), Orange, California
  - UC Irvine Health ( Site 0029), Orange, California
  - Providence Saint John's Health Center ( Site 0083), Santa Monica, California
  - Georgetown University Medical Center ( Site 0006), Washington D.C., District of Columbia
  - AdventHealth Orlando-AdventHealth Medical Group Hematology & Oncology at Orlando ( Site 0003), Orlando, Florida
  - Orlando Health, Inc. ( Site 0035), Orlando, Florida
  - University Cancer & Blood Center, LLC ( Site 0057), Athens, Georgia
  - Emory University Hospital ( Site 0012), Atlanta, Georgia
  - Rush University Medical Center ( Site 0040), Chicago, Illinois
  - Illinois Cancer Care, PC ( Site 0008), Peoria, Illinois
  - Parkview Cancer Institute ( Site 0088), Fort Wayne, Indiana
  - Norton Cancer Institute - St. Matthews ( Site 0065), Louisville, Kentucky
  - Tulane University School of Medicine ( Site 0098), New Orleans, Louisiana
  - Lahey Hospital & Medical Center ( Site 0090), Burlington, Massachusetts
  - Cancer & Hematology Centers of Western Michigan ( Site 0018), Grand Rapids, Michigan
  - HealthPartners Cancer Research Center-HealthPartners Frauenshuh Cancer Center ( Site 0005), Saint Louis Park, Minnesota
  - University of Mississippi Medical Ctr ( Site 0037), Jackson, Mississippi
  - Cancer Partners of Nebraska ( Site 0086), Lincoln, Nebraska
  - Rutgers Cancer Institute of New Jersey ( Site 0078), New Brunswick, New Jersey
  - R.J. Zuckerberg Cancer Center-Medical Oncology ( Site 0013), Lake Success, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0055), New York, New York
  - Levine Cancer Institute ( Site 0004), Charlotte, North Carolina
  - Duke Cancer Institute ( Site 0096), Durham, North Carolina
  - Lehigh Valley Hospital- Cedar Crest-Oncology Clinical Trials ( Site 0056), Allentown, Pennsylvania
  - University of Texas, Southwestern Medical Center ( Site 0015), Dallas, Texas
  - Huntsman Cancer Institute-HCI Clinical Trials Office ( Site 7001), Salt Lake City, Utah
  - University of Vermont Medical Center ( Site 0001), Burlington, Vermont
  - Blue Ridge Cancer Care - Roanoke ( Site 0043), Roanoke, Virginia
  - Seattle Cancer Care Alliance-Renal/Melanoma/MCC ( Site 0093), Seattle, Washington
  - Confluence Health | Wenatchee Valley Hospital & Clinics ( Site 0061), Wenatchee, Washington
- Argentina (6):
  - Centro de Urología (CDU) ( Site 0803), CABA, Buenos Aires
  - Hospital Británico de Buenos Aires-Oncology ( Site 0801), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming ( Site 0800), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Sanatorio Británico-Clinical Oncology Department ( Site 0802), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 0806), Rosario, Santa Fe Province
  - Asociación de Beneficencia Hospital Sirio Libanés ( Site 0804), Buenos Aires
- Australia (4):
  - GenesisCare North Shore ( Site 4011), St Leonards, New South Wales
  - Lyell McEwin Hospital ( Site 4004), Elizabeth Vale, South Australia
  - Peninsula Health Frankston Hospital ( Site 4001), Frankston, Victoria
  - Peter MacCallum Cancer Centre-Parkville Cancer Clinical Trials Unit (PCCTU) ( Site 4010), Melbourne, Victoria
- Austria (5):
  - Medizinische Universitätsklinik Graz ( Site 1051), Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen-Urologie ( Site 1001), Linz, Upper Austria
  - Klinik Ottakring-1.Medizinische Abteilung - Zentrum für Onkologie und Hämatologie ( Site 1031), Vienna, Vienna
  - Krankenhaus der Barmherzigen Brüder Wien ( Site 1041), Vienna
  - Medizinische Universität Wien ( Site 1021), Vienna
- Belgium (6):
  - Institut Jules Bordet ( Site 1103), Anderlecht, Bruxelles-Capitale, Region de
  - Cliniques Universitaires Saint Luc - Bruxelles ( Site 1105), Brussels, Bruxelles-Capitale, Region de
  - Grand Hopital de Charleroi ( Site 1104), Charleroi, Hainaut
  - UZ Gent ( Site 1100), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 1101), Leuven, Vlaams-Brabant
  - CHU de Liege ( Site 1102), Liège
- Brazil (4):
  - Liga Norte Riograndense Contra o Cancer ( Site 0313), Natal, Rio Grande do Norte
  - Centro Gaucho Integrado de Oncologia ( Site 0304), Porto Alegre, Rio Grande do Sul
  - BP - A Beneficencia Portuguesa de São Paulo-Medical Oncology ( Site 0311), São Paulo
  - Hospital Paulistano - Amil Clinical Research ( Site 0308), São Paulo
- Canada (11):
  - Tom Baker Cancer Centre ( Site 0109), Calgary, Alberta
  - Cross Cancer Institute ( Site 0111), Edmonton, Alberta
  - BC Cancer Vancouver-Clinical Trials Unit ( Site 0110), Vancouver, British Columbia
  - The Moncton Hospital ( Site 0101), Moncton, New Brunswick
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0114), Hamilton, Ontario
  - Kingston Health Sciences Centre ( Site 0105), Kingston, Ontario
  - The Ottawa Hospital - General Campus-The Ottawa Hospital Cancer Centre ( Site 0116), Ottawa, Ontario
  - Sunnybrook Health Sciences - Odette Cancer Centre ( Site 0113), Toronto, Ontario
  - CISSS de la Monteregie-Centre ( Site 0103), Greenfield Park, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0102), Sherbrooke, Quebec
- Chile (2):
  - Bradfordhill-Clinical Area ( Site 0400), Santiago, Region M. de Santiago
  - James Lind Centro de Investigación del Cáncer ( Site 0402), Temuco, Región de la Araucanía
- Colombia (4):
  - Fundación Colombiana de Cancerología Clínica Vida ( Site 0505), Medellín, Antioquia
  - Sociedad De Oncologia Y Hematologia Del Cesar-Oncology ( Site 0508), Valledupar, Cesar Department
  - Instituto Nacional de Cancerología-Clinical Oncology ( Site 0500), Bogotá, Cundinamarca
  - Fundación Cardiovascular de Colombia ( Site 0501), Piedecuesta, Santander Department
- Czechia (5):
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 2203), Brno, Brno-mesto
  - Nemocnice České Budějovice-Onkologicke oddeleni ( Site 2204), České Budějovice, Jihočeský kraj
  - Fakultni Thomayerova nemocnice-Onkologicka klinika 1. LF UK ( Site 2200), Prague, Praha 4
  - Fakultni nemocnice v Motole-Onkologicka klinika 2. LF UK a FN Motol ( Site 2205), Prague, Praha 5
  - Fakultni nemocnice Hradec Kralove-Klinika onkologie a radioterapie ( Site 2201), Hradec Králové
- Finland (3):
  - Tampereen yliopistollinen sairaala ( Site 1801), Tampere, Pirkanmaa
  - TYKS ( Site 1802), Turku, Southwest Finland
  - HYKS ( Site 1800), Helsinki, Uusimaa
- France (9):
  - Institut Jean Godinot ( Site 1216), Reims, Ain
  - Centre Antoine Lacassagne ( Site 1217), Nice, Alpes-Maritimes
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 1218), Strasbourg, Alsace
  - CHU de Bordeaux- Hopital Saint Andre ( Site 1209), Bordeaux, Gironde
  - Institut Claudius Regaud ( Site 1215), Toulouse, Haute-Garonne
  - Clinique Francois Chenieux ( Site 1210), Limoges, Haute-Vienne
  - Institut de Cancerologie de l Ouest Centre Rene Gauducheau ( Site 1201), Saint-Herblain, Loire-Atlantique
  - Institut de Cancerologie de l Ouest Site Paul Papin ( Site 1200), Angers, Maine-et-Loire
  - Hopital Tenon ( Site 1213), Paris
- Germany (10):
  - Klinik fuer Urologie ( Site 1303), Freiburg im Breisgau, Baden-Wurttemberg
  - NCT-Department of Medical Oncology ( Site 1320), Heidelberg, Baden-Wurttemberg
  - Klinikum Nuernberg Nord ( Site 1300), Nuremberg, Bavaria
  - Universitaetsklinikum Frankfurt ( Site 1301), Frankfurt am Main, Hesse
  - Universitaetsklinikum Aachen AOER ( Site 1317), Aachen, North Rhine-Westphalia
  - Universitaetsklinikum des Saarlandes ( Site 1305), Homburg/ Saar, Saarland
  - Krankenhaus Martha Maria Halle-Doelau ( Site 1314), Halle, Saxony-Anhalt
  - Helios Klinikum Erfurt GmbH ( Site 1315), Erfurt, Thuringia
  - Charite Universitaetsmedizin Berlin ( Site 1321), Berlin
  - HELIOS Klinikum Berlin-Buch ( Site 1311), Berlin
- Greece (5):
  - UNIVERSITY HOSPITAL OF PATRAS-DIVISION OF ONCOLOGY ( Site 3302), Pátrai, Achaia
  - Alexandra General Hospital of Athens-ONCOLOGY DEPT. ( Site 3304), Athens, Attica
  - Athens Medical Center ( Site 3303), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL ( Site 3301), Chaïdári, Attica
  - European Interbalkan Medical Center-Oncology Department ( Site 3300), Thessaloniki
- Ireland (3):
  - Mater Misericordiae University Hospital ( Site 3201), Dublin, Dublin
  - Tallaght University Hospital ( Site 3200), Dublin
  - Mater Private Hospital - Dublin ( Site 3202), Dublin
- Italy (11):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori ( Site 1407), Meldola, Forli-Cesena
  - Istituto Clinico Humanitas Research Hospital ( Site 1406), Rozzano, Milano
  - Ospedale San Luigi Gonzaga ( Site 1405), Orbassano, Torino
  - Medical Oncology Ospedale San Donato ( Site 1404), Arezzo
  - Azienda Ospedaliera Policlinico di Bari ( Site 1402), Bari
  - IRCCS Ospedale San Raffaele ( Site 1409), Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 1400), Milan
  - Istituti Clinici Scientifici Maugeri Spa ( Site 1403), Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli-Medical Oncology ( Site 1410), Roma
  - Azienda Ospedaliera S. Maria di Terni ( Site 1401), Terni
  - Ospedale Maggiore Borgo Trento ( Site 1408), Verona
- Japan (18):
  - Fujita Health University ( Site 5003), Toyoake, Aichi-ken
  - National Cancer Center Hospital East ( Site 5000), Kashiwa, Chiba
  - Toho University Sakura Medical Center ( Site 5014), Sakura, Chiba
  - Sapporo Medical University Hospital ( Site 5008), Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital ( Site 5017), Kobe, Hyōgo
  - Yokohama City University Hospital ( Site 5007), Yokohama, Kanagawa
  - Nara Medical University Hospital ( Site 5002), Kashihara, Nara
  - Kindai University Hospital- Osakasayama Campus-Urology ( Site 5010), Sayama, Osaka
  - Osaka University Hospital ( Site 5012), Suita, Osaka
  - Hamamatsu University School of Medicine University Hospital ( Site 5004), Hamamatsu, Shizuoka
  - Tokyo Medical and Dental University Hospital ( Site 5009), Bunkyo-ku, Tokyo
  - Toranomon Hospital ( Site 5001), Minato-ku, Tokyo
  - Kyushu University Hospital ( Site 5005), Fukuoka
  - Niigata University Medical & Dental Hospital ( Site 5013), Niigata
  - Osaka International Cancer Institute ( Site 5016), Osaka
  - Nippon Medical School Hospital ( Site 5006), Tokyo
  - Tokyo Women's Medical University Adachi Medical Center ( Site 5015), Tokyo
  - Keio university hospital ( Site 5011), Tokyo
- Netherlands (8):
  - Zuyderland Medical Centre-Trialbureau Interne Geneeskunde ( Site 1904), Sittard-Geleen, Limburg
  - Amphia Hospital Location Molengracht ( Site 1912), Breda, North Brabant
  - Antoni van Leeuwenhoek Ziekenhuis ( Site 1901), Amsterdam, North Holland
  - Medisch Centrum Leeuwarden ( Site 1905), Leeuwarden, Provincie Friesland
  - Erasmus MC ( Site 1913), Rotterdam, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Vlietland ( Site 1909), Schiedam, South Holland
  - Haga Ziekenhuis locatie Leyweg-Oncology ( Site 1917), The Hague, South Holland
  - Universitair Medisch Centrum Utrecht ( Site 1910), Utrecht
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Poznaniu ( Site 2401), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 2402), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - O-Klinika Onkologii Klinicznej ( Site 240, Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 2400), Warsaw, Masovian Voivodeship
- Romania (3):
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 2500), Cluj-Napoca, Cluj
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 2501), Cluj-Napoca, Cluj
  - Centrul de Oncologie "Sfântul Nectarie" ( Site 2502), Craiova, Dolj
- Russia (7):
  - Ivanovo Regional Oncology Dispensary ( Site 2616), Ivanovo, Ivanovo Oblast
  - FSBI United Hospital with Polyclinic ( Site 2613), Moscow, Moscow
  - SHI of Moscow City Oncology Clinical Hospital - 62 ( Site 2614), Moscow, Moscow
  - MEDSI Clinical Hospital on Pyatnitsky Highway-Departmentof Antitumor Drug therapy ( Site 2618), Krasnogorsk, Moscow Oblast
  - Hadassah Medical-Oncology department ( Site 2609), Moscow, Moscow Oblast
  - Volgograd Regional Uronephrological Center ( Site 2615), Volzhsky, Volgograd Oblast
  - Yaroslavl Regional Cancer Hospital-Oncology ( Site 2619), Yaroslavl, Yaroslavl Oblast
- South Korea (3):
  - Chonnam National University Hwasun Hospital-Oncology ( Site 4203), Hwasun, Jeonranamdo
  - Asan Medical Center ( Site 4200), Seoul
  - Samsung Medical Center ( Site 4201), Seoul
- Spain (8):
  - Complejo Hospitalario Universitario A Coruna ( Site 1502), A Coruña, La Coruna
  - Hospital Universitario 12 de Octubre-Medical Oncology ( Site 1508), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 1507), Barcelona
  - Hospital Clinic i Provincial ( Site 1500), Barcelona
  - Hospital Santa Creu i Sant Pau ( Site 1501), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 1505), Madrid
  - Hospital Clinico San Carlos ( Site 1504), Madrid
  - Hospital Virgen del Rocio ( Site 1503), Seville
- Switzerland (4):
  - Hopitaux Universitaires de Geneve HUG ( Site 1602), Geneva, Canton of Geneva
  - Universitaetsspital Zuerich ( Site 1601), Zurich, Canton of Zurich
  - Istituto Oncologica della Svizzera Italiana (IOSI) ( Site 1604), Bellinzona, Canton Ticino
  - Kantonsspital Graubuenden ( Site 1600), Chur, Kanton Graubünden
- United Kingdom (8):
  - Aberdeen Royal Infirmary-Department of Oncology ( Site 3105), Aberdeen, Aberdeen City
  - Royal United Hospital Bath England ( Site 3108), Bath, Bath And North East Somerset
  - Nottingham University Hospitals NHS Trust. City Hospital Campus ( Site 3106), Nottingham, England
  - Southend University Hospital ( Site 3112), Southend, Essex
  - Imperial Healthcare NHS Trust Charing Cross Hospital ( Site 3107), London, London, City of
  - Mount Vernon Cancer Centre ( Site 3101), Northwood, London, City of
  - Musgrove Park Hospital ( Site 3103), Taunton, Somerset
  - Singleton Hospital ( Site 3111), Swansea, Wales

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Motzer RJ, Schmidinger M, Eto M, Suarez C, Figlin R, Liu Y, Perini R, Zhang Y, Heng DY. LITESPARK-011: belzutifan plus lenvatinib vs cabozantinib in advanced renal cell carcinoma after anti-PD-1/PD-L1 therapy. Future Oncol. 2023 Jan;19(2):113-121. doi: 10.2217/fon-2022-0802. Epub 2023 Feb 8. PMID 36752726
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26229&tenant=MT_MSD_9011